CLINICAL TRIAL: NCT03201328
Title: Prospective, Single Centre Cohort Study on the Impact of Binaural Audition on Postural Performance and Orientation in Healthy Subjects and Patients With Cochlear Implants.
Brief Title: Impact of Binaural Audition on Postural Performance and Orientation
Acronym: AUDIPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOZORG GRAYELI GUIGOU UB 2015
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Unilateral Cochlear Implants; Bilateral Cochlear Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy subjects (Active Comparator)
  Interventions: Other: Audio-vestibular examination; Other: Videonystagmoscopic study; Other: Posturographies study
- patients with unilateral cochlear implants (Experimental)
  Interventions: Other: Audio-vestibular examination; Other: Videonystagmoscopic study; Other: Posturographies study
- patients with bilateral cochlear implants (Experimental)
  Interventions: Other: Audio-vestibular examination; Other: Videonystagmoscopic study; Other: Posturographies study

INTERVENTIONS:
Other: Audio-vestibular examination — Vestibular tests (videonystagmoscopy and head video impulse test), the tonal and vocal audiogram and the localigramme to the cochlear implanted subjects. Tonal audiometry and localigramme to the healthy subjects.
Other: Videonystagmoscopic study — Rotating sound stimulation on a rotatory armchair and a laborer of Fukuda with sound stimulation and questionary before and after examination.
Other: Posturographies study — (stabilometry, sensory preferences, indications of energy consumption) with stereophonic stimulation and questionnaire before and after the examination.

SUMMARY:
This is a prospective research study talking place at University hospital of Dijon and requiring the inclusion of 20 healthy subjects, 10 patients with unilateral cochlear implants and 10 patients with bilateral cochlear implants to carry out:

* an audio-vestibular examination,
* a videonystagmoscopic study,
* a posturography study and
* a movement study. The aim of the study is to evaluate the impact of binaural audition on postural performance and orientation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written consent
* Patients with health insurance cover
* Age between 18 and 75 years old
* For subjects with implants: unilateral or bilateral cochlear implants for more than one year
* For healthy subjects: absence of known audio-vestibular disorders (deafness, vertigo)

Exclusion Criteria:

* Patients dependent on an aid to move around (cane, wheelchair, crutch, ...)
* Patients under guardianship
* Pregnant women
* Disability interfering with understanding or carrying out instructions
* Associated sensory or motor disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Presence of a sensation of rotation due to a turning sound source | Baseline
Modification of posturography parameters in the presence and absence of a de turning sound source | Baseline
Time to cover a distance of 3metres in a straight line and number of steps used | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France